CLINICAL TRIAL: NCT00834535
Title: A Relative Bioavailability Study of 300 mg Cefdinir Capsules Under Non-fasting Conditions
Brief Title: Cefdinir Capsules 300 mg, Non-fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R04-1123
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Cefdinir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cefdinir Capsules 300 mg
- 2 (Active Comparator)
  Interventions: Drug: OMNICEF® Capsule 300 mg

INTERVENTIONS:
Drug: Cefdinir Capsules 300 mg — 1 x 300 mg, single-dose non-fasting
  Arms: 1
Drug: OMNICEF® Capsule 300 mg — 1 x 300 mg, single-dose non-fasting
  Arms: 2

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 300 mg Cefdinir Capsules manufactured and distributed by TEVA pharmaceuticals USA with that of OMNICEF® Capsules by CEPH International Corporation for Abbott Laboratories following a single oral dose (1 x 300mg capsule) in healthy adult subjects administered under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All subjects selected for this study will be healthy men and women 18 years of age or older at the time of dosing. the subject's body mass index (BMI) should be 19 kg/m² - 30 kg/m², inclusive.
* Screening procedures: Each subject will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems.

The screening clinical laboratory procedures will include:

* Hematology: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count;
* Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
* HIV antibody and hepatitis B surface antigen and hepatitis C antibody screens;
* Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
* Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
* Serum Pregnancy Screen (female subjects only)

If female and:

* of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condom with spermicide, diaphragm with spermicide, intrauterine device (IUD) or abstinence; or
* is postmenopausal for at least 1 year; or
* is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Subjects with a recent history of drug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody or HIV antibody.
* Subjects demonstrating a positive drug abuse screen when screened for this study.
* Female subjects demonstrating a positive pregnancy screening.
* Female subjects who are currently breastfeeding.
* Subjects with a history of allergic response(s) to cefdinir or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently use or report using tobacco products within 3 months of Period I dose administration.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subjects who have donated serum (e.g. serumpheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate serum for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.
* Subjects who report having difficulty fasting or consuming standardized meals.
* Female subjects who report using implanted or injected hormonal contraceptives (birth control) during the 6 months prior to Period I dosing.
* Female subjects who report using oral hormonal contraceptives (birth control) during the 14 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (2):
- United States (2):
  - PRACS Institute, Ltd., East Grand Forks, Minnesota
  - PRACS Institute, Ltd., Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefdinir (Test) First: 300 mg Cefdinir Capsules test product dosed in first period followed by 300 mg Omnicef® Capsules reference product dosed in the second period.
- Omnicef® (Reference) First: 300 mg Omnicef® Capsules reference product dosed in first period followed by 300 mg Cefdinir Capsules test product dosed in the second period.
Period: First Intervention
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 14 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cefdinir (Test): 300 mg Cefdinir Capsules test product dosed in either period.
- Omnicef® (Reference): 300 mg Omnicef® Capsules reference product dosed in either period.
Arm/Group | Cefdinir (Test) | Omnicef® (Reference)
Number analyzed (Participants) | 32 | 32
ng/mL | 2081.37 (537.12) | 2045.43 (481.25)
Statistical Analysis 1: Comparison: Cefdinir (Test) vs Omnicef® (Reference); Test type: Non-Inferiority or Equivalence — The ANOVA model containing factors for sequence of products, subjects within sequence, periods, and products was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 100.83, 90% CI [93.98 to 108.17] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 14 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefdinir (Test) | Omnicef® (Reference)
Number analyzed (Participants) | 32 | 32
ng*h/mL | 10700.97 (2328.12) | 11121.51 (2215.78)
Statistical Analysis 1: Comparison: Cefdinir (Test) vs Omnicef® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 96.1, 90% CI [92.14 to 100.22] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 14 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefdinir (Test) | Omnicef® (Reference)
Number analyzed (Participants) | 32 | 32
ng*h/mL | 11219.51 (2304.28) | 11560.85 (2237.52)
Statistical Analysis 1: Comparison: Cefdinir (Test) vs Omnicef® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 96.57, 90% CI [92.8 to 100.49] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.